CLINICAL TRIAL: NCT07045493
Title: Assessing Safety and Efficacy of Ivermectin and Albendazole Combination Therapy for Soil-transmitted Helminthiasis in Pre-school-aged Children (PSAC) in Bangladesh
Brief Title: Assessing the Safety and Efficacy of a Combination Therapy for STH in PSAC in Bangladesh
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Cures Within Reach (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR-25009
Record Dates: First submitted 2025-04-27; First posted 2025-07-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Soil Transmitted Helminth (STH) Infections
MeSH Terms: conditions — Infections | interventions — Albendazole; Ivermectin; Combined Modality Therapy

STUDY DESIGN:
Intervention Model Description: This will be a Phase IIa, single-blinded, clinical superiority, randomized controlled trial where the safety and efficacy of ivermectin and albendazole combination therapy will be evaluated compared to the standard medication (albendazole monotherapy) against soil-transmitted helminths amongst the preschool-aged children aged between 2 and 5 years.
Who Masked: Outcomes Assessor
Masking Description: This study will be a single-blinded clinical trial. The investigators and study physicians will not be blinded. The investigators are not using any placebo arm for this trial; the approach to concealing the treatment arm by random selection of the study participants will avoid selection bias in the study. However, the primary objective of the study is a cure assessment of STH infection, which will be performed based on the egg reduction rate (ERR) with stool samples. To ensure the avoidance of any bias in the test, the laboratory personnel doing the procedures will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm - 1 (Experimental): A single dose of Albendazole 400mg + Ivermectin (200 µg/kg) combination therapy
  Interventions: Drug: A single dose of Albendazole 400mg + Ivermectin (200 µg/ kg) combination therapy
- Treatment Arm - 2 (Active Comparator): A single dose of 400 mg Oral Albendazole monotherapy
  Interventions: Drug: A single dose of 400 mg Oral Albendazole monotherapy

INTERVENTIONS:
Drug: A single dose of Albendazole 400mg + Ivermectin (200 µg/ kg) combination therapy — Children will receive the medication after being randomly assigned to either treatment arm. Albendazole will be administered as a syrup and ivermectin tablets as powdered tablets because ivermectin suspension is not available in Bangladesh. The commercially available 6 mg unscored Ivermectin tablets will be crushed, the tablet fragments ground into a powder, and stored in an airtight plastic container in a dry, cool environment after all aseptic procedures. According to the weight of the children, the investigators will provide the needed amount (weighted by microgram scale) of the drug mixed with 5 ml of water. The study field staff will help the parents to give the medicine to the child by the direct observation therapy (DOT) method. The parents will be advised to bring the children on an empty stomach in the morning. Ivermectin will be given first, and a light snack will be provided 30 minutes after taking ivermectin. Then albendazole will be given to the children.
  Arms: Treatment Arm - 1
Drug: A single dose of 400 mg Oral Albendazole monotherapy — Albendazole will be given in syrup form. The study field staff will help the parents to give the medicine to the child by the direct observation therapy (DOT) method. The parents will be advised to bring the children on an empty stomach in the morning. Ivermectin will be given first, and a light snack will be provided 30 minutes after taking ivermectin. Then albendazole will be given to the children. Both drugs will be given using direct observation at the field clinic. Parents will be advised to report any adverse effects, including vomiting, after taking the medication. If vomiting occurs within one hour of medication, a redosing will be provided.
  Arms: Treatment Arm - 2

SUMMARY:
Background (brief):

1. Burden:

   Soil-transmitted helminth (STH) infections are a major public health problem, primarily affecting children. Although STH prevalence has decreased to 14% in Bangladesh, over 47 million preschool- and school-age children still live in high-risk areas.
2. Knowledge gap:

   Albendazole shows 94-100% efficacy against A. lumbricoides but only 39-60% against T. trichuria. Ivermectin is also effective against hookworm and T. trichuria. Combining ivermectin with albendazole may be more effective than using either drug alone, but this combined therapy for STH has not yet been studied in Bangladesh.
3. Relevance:

STHs significantly impact children's nutrition, hindering health, growth, cognition, and learning. The national deworming program achieved 98.3% treatment coverage, but only 76.2% of PSAC were dewormed using self-prescribed medicines.

Hypothesis (if any):

The combination therapy of Albendazole and Ivermectin is more effective than Albendazole alone for treating soil-transmitted helminths in preschool-age children in Bangladesh

Objectives:

1. To compare the safety and efficacy of Albendazole and Ivermectin combination therapy with Albendazole monotherapy in preschool-aged children
2. To evaluate post-treatment egg reduction rates for various helminths at different time points
3. To determine the median time to re-infection following different anti-helminth interventions for various STH

Methods:

This Phase IIa single-blinded, randomized controlled trial will evaluate the safety and efficacy of ivermectin and albendazole combination therapy versus standard albendazole monotherapy for STH in 2-5 years in rural Belkuchi, Sirajganj. A total of 110 PSAC with confirmed STH will be randomly assigned to two treatment arms. Field activities and laboratory analysis will use the Kato-Katz technique for microscopic examination.

Outcome measures/variables:

* Evaluate the safety and efficacy of ivermectin and albendazole combination therapy for STH
* Evaluate the statistically significant impact on patient clinical outcomes, cure rate, and egg reduction rate
* Correlate changes in Cure Rate and Egg Reduction Rate for different STH at various time points

DETAILED DESCRIPTION:
Description of the Research Project

Background of the Project including Preliminary Observations:

Epidemiology of Soil-transmitted helminthiasis Soil-transmitted helminthiasis (STH) infections are a group of parasitic infections caused by Ascaris lumbricoides (AL), Trichuris trichiura (TT), Ancylostoma duodenale (AD) and Necator americanus (NA) (hookworms). This infection is transmitted to humans by contaminated soil by human faeces containing parasite eggs. These infections impact the most impoverished and marginalized communities that lack access to clean water, sanitation, and proper hygiene, particularly in tropical and subtropical regions. At the same time, the highest prevalence is documented in sub-Saharan Africa, China, South America, and Asia. STH is a significant public health threat, with an estimated 1.5 billion people or 24% of the world population resulting in a loss of two million disability-adjusted life years.

The nutritional status of STH-infected children is often affected, eventually leading to impaired health, growth, cognition, and educational outcomes. High helminth intensity and polyparasitism may cause malnourishment and morbidity, which may result in death. Because of physical barrier and/or competition for food, helminths may make human hosts' malnutrition worse. Insufficient absorption of micronutrients and intestinal blood loss are more intricately linked to anaemia through an unknown process. The overall effect may change the children's cognitive development, including memory, reaction time, learning, and intrinsic intelligence. Children in preschool are not currently included in regular deworming programs for STH. However, the research indicates that children get infected soon after weaning and continue to be infected throughout childhood and adolescence. Children are negatively impacted by infections long before attending school, which exacerbates the long-term health risks of STH infection. Epidemiological research conducted among SACs demonstrated that STHs had a direct impact on student performance and absenteeism. So, deworming may play vital roles for preschool-aged children before entering school.

Several demographic groups are considered eligible for routine deworming, including preschool-aged children (PSAC) and school-aged children (SAC). In Bangladesh, STH was prevalent among 79.8% of school-age children (SAC) in 2005, which dropped to 14% in recent times. The prevalence is higher in slums or low socio-economic clusters (around 50.54%) due to poor hygiene and malnutrition, despite homogenous mass drug administration, MDA. More than one-third (36.3%) of SAC are re-infected with at least one helminth within six months of the MDA, with the highest prevalence of TT (27.5%) and 12.4 % of multiple helminth infections, which indicates the inefficiency of current PC.

Bangladesh Ministry of Health & Family Welfare (MOHFW) and Children Without Worms (CWW) conducted the Integrated Community-based Survey for Program Monitoring" (ICSPM) in 4 districts in 2016 and 10 districts from 2017-2020. According to both surveys, the moderate-to-high intensity infection of STH (MHII) was one of the highest in Sirajganj (7.1%) and it was above the WHO-recommended target of <1%. A. lumbricoides was the most common STH parasite followed by T. trichiura and hookworm. A. lumbricoides was most prevalent among SAC (n = 139,8.9% ), followed by PSAC (n = 114, 8.1% ) and adults n = 99, 7.4%,). All polyparasitism was due to A. lumbricoides and T. trichiura (n = 14,0.3% ) and was only identified in Sirajganj District. Sirajganj subdistricts of concern included Belkuchi (STH prevalence in SAC: 57.1%, 20.0% MHII) and Kamarkhanda (STH prevalence in SAC: 50.0%, 28.6% MHII). Belkuchi had the highest STH prevalence in PSAC (n = 23, 60.5% ), SAC (n = 20, 57.1% ), and adults (n = 15, 50.0% ). Belkuchi had the highest MHII among PSAC [(n = 9, 23.7%) and adults (n = 6, 20.0%), and Kamarkhanda had the highest MHII among SAC.

Treatment of STH- Bangladesh perspective The latest WHO roadmap for neglected tropical diseases aims to eliminate STHs as a public health concern in 96% of endemic countries by 2030. To combat STH the WHO suggests four medications for treating STH infections: pyrantel, levamisole, mebendazole, and albendazole. WHO introduced routine preventive chemotherapy (PC) for preschool and school-aged children, using benzimidazoles (albendazole or mebendazole) in 2001. The benzimidazole medications, such as albendazole and mebendazole, work by disrupting the parasitic worms' microtubular system to treat a range of parasitic infections. These are the most common medications used to treat roundworm and hookworm. These are inexpensive, secure, and simple to use as children do not need to be weighed. Both adults and children receive the same dosage. However, Albendazole and mebendazole, commonly dispensed against soil-transmitted helminths (STH), are frequently utilized in combination with other medications to establish an integrated approach.

The widespread use of these medications for treatment and preventative chemotherapy is a result of the excellent efficacy demonstrated by the applications of scientific knowledge. Through WHO, national health ministries in endemic countries get donations of albendazole and mebendazole to treat school-age children. Bangladesh implemented a national deworming program in 2008, which involves MDA at primary schools for age groups 6-12 years with Mebendazole/Albendazole (ALB) monotherapy as preventive chemotherapy (PC), conducted at six-month intervals. The deworming program had reached a national treatment coverage increasing from 86.4% to 98.3% in the four years 2015-2019; however, only 76.2% of PSAC were found to be dewormed through self-prescribed locally purchased deworming medicines.

Current Treatment Review Since 1982, Albendazole has been used extensively to treat intestinal parasites. High cure rates for lumbricoides infections are attained with a single dosage of albendazole. The cure rates attained in various trials, however, vary. The efficacy of ALB against AL infection is well established with a 94%-100% egg reduction rate (ERR), while it has proved inefficient in curbing TT infections (ERR: 39%-60%). A single oral dose of albendazole, mebendazole, and pyrantel pamoate effectively treats infections caused by Ascaris lumbricoides, but a single dose of mebendazole was ineffective in combating hookworm infections in school children in Zanzibar and Vietnam. A quick re-infection, especially in the case of AL and TT, was found in another study aiming to assess patterns and dynamics of STH reinfection after drug treatment. However, treating infections from Trichuris trichiura with the current anthelmintics in a single oral dose is unsatisfactory. The side effects of albendazole include headache, leukopenia, and temporary gastrointestinal distress.

Scope of Repurposing Ivermectin in STH Ivermectin (IVM) is a safe and widely used macrocyclic lactone due to its broad-spectrum anti-infective and anti-parasitic activity against ecto- and endoparasites. Ivermectin is mostly used to treat strongyloidiasis, loiasis, onchocerciasis, and lymphatic filariasis. Additionally, it has been licensed to treat human ascariasis and has a beneficial effect on Trichuris trichiura. It paralyzes adult worms and appears to be dormant. Indirect evidence suggests a decreased burden of soil-transmitted helminths in regions where albendazole and ivermectin have been jointly administered. While ivermectin alone is recognized for having less-than-optimal efficacy against hookworm and TT infections, available data indicates that the combined administration of ivermectin and albendazole may exhibit greater efficacy compared to single-drug regimens. The co-administration of ivermectin and albendazole significantly outperformed albendazole alone in clearing TT infections, with a relative risk (RR) of 0.44 (95% CI = 0.31-0.62) for post-treatment infection. Patients receiving the combination treatment demonstrated higher individual egg reduction rates (ERRs) ranging from 91% to 100%, a cumulative cure rate (CR) of 45.8%, and an overall ERR of 84.5%, surpassing the efficacy of albendazole alone (ERR = 59.1%) and Ivermectin alone (ERR = 72.1%) (p < 0.001). Ivermectin-treated patients have not seen any significant side effects, according to safety trials. Adverse effects of ivermectin included abdominal pain, headache, and diarrhoea .

Relevance for assessing new treatment regimen The two benzimidazole medications mebendazole (500 mg) and albendazole (400 mg) are currently used primarily to treat STH infections. Both medications are highly effective against A. lumbricoides (cure rate (CR) = 96% with albendazole and CR = 96% with mebendazole), according to a 2017 meta-analysis. However, these are less effective against hookworm (CR = 80% with albendazole and CR = 33% with mebendazole), and less effective against T. trichiura (CR = 31% with albendazole and CR = 42% with mebendazole). Given the enormous drug pressure imposed by widespread usage and dependence on these two medications, it is imperative to step up efforts to investigate alternative medicines to both improve efficacy for trichuriasis and postpone the establishment of potential drug resistance.

In regions where albendazole and ivermectin have been co-administered, there is indirect evidence of a lower burden of STH. Data suggests that ivermectin and albendazole administered together can be more effective than single-drug regimens, even though ivermectin alone is thought to have inadequate efficacy against hookworm and T. trichiura infections . As a result, the WHO Essential Medicines List now includes ivermectin and albendazole together for the treatment of STH infection. Future MDA campaigns are expected to support the use of ivermectin-albendazole co-treatment since it is listed in the WHO Model List of Essential Medicines to treat STH.

As the WHO suggested revising the frequency of MDA treatments, the discovery of therapy to increase efficacy, delay the reinfection time, and halt the emergence of potential drug resistance is paramount. Evidence does exist that PSAC benefits from deworming, and others have advocated for PSAC inclusion in MDA. Deworming of PSAC will help to address the infections at the earlier stages, potentially preventing the progression of disease and associated complications. Besides that, the upscaling of PC over the past years has increased the selective drug pressure on STH-affected populations, posing the risk of triggering anthelmintic drug resistance. In addition, deworming PSAC complements efforts to break the cycle of transmission within communities, reducing the overall burden of STH infections.

Research Design and Methods

Research plan/experimental design:

Study Site The research will be conducted in rural settings in the Belkuchi sub-district (upazila) of Sirajganj district, which had the highest STH prevalence among PSACs (60.5%). The investigators will set up a field office there for conducting patient screening, enrolment, microscopic examination, treatment, and follow-up.

Study Population In this study, the investigators will screen about 300 preschool-aged children (PSAC) by household visits to the study site, and then the investigators will randomly select 110 pre-SACs following all the inclusion and exclusion criteria and put them into randomization for selecting treatment arm.

Screening and enrolment of the patients:

The study will be done in a rural area (Belkuchi Sub-district) of Sirajganj District of Bangladesh. The investigators will set up a field office in the study area with a radius of about 5 km from the office. At the initiation phase of the project, a household (HH) survey will be conducted in the study area after obtaining consent from the HH head(s). Trained field assistants will visit every house of the study site and enlist children falling within the age limit. Parents or guardians of the enlisted children will be invited and will receive detailed information about the study's objectives, procedures, potential benefits, and risks. The investigators will hold an open discussion session encouraging parents and others to ask questions and provide ample time for them to decide whether to allow the children to participate. Then, the investigators will obtain informed written consent from parents or guardians of the eligible children. At baseline, the study physician, the medical lab technician, and trained field assistants will be assigned to screen the participants and collect stool samples from potential participants for examination for STH. Participants will be enrolled in compliance with the study inclusion and exclusion criteria after being examined by the study physician to ensure maximum patient safety. All the study activities, including the participant screening, will be done after the proper consent of the parents / legal guardians of the participants. The investigators will document the details of all eligible children, including name, sex, age, and school grade. Then the investigators will ask them for having any clinical symptoms and perform physical examinations. Additionally, The investigators will measure height to the nearest centimetres, and weight will be recorded to the nearest 0.1 kg. A sterile empty stool container will be provided to the parents of eligible children, marked with unique identification numbers, and parents will be asked to return the container along with a fresh morning stool sample of the child.

Treatment Allocation:

The enrolled participants will be randomly assigned to one of the treatment arms through individual randomization using MS Excel software. Each patient will draw a sealed and numbered envelope and thus have an equal chance to receive either of the regimens. The investigators will not use block randomization. As the study participants are 2-5 years old and the investigators will conduct the study on a single site, the investigators will use open randomization using numbered envelopes. Treatment Regimen will be assigned a random number 1-110, 55 in each arm. Inside the chosen envelope there will be a card specifying the assigned treatment - either the "Standard Treatment Regimen" (Albendazole 400mg monotherapy) or the "Combination Therapy Treatment Regimen" (a single dose of Albendazole 400mg + Ivermectin (200 μg/kg). The selected card is then placed back into the envelope for drug accountability and monitoring purposes. The approach to concealing the treatment arm by random selection of the study participants will avoid selection bias in the study.

Drug Dispensing:

After being randomized to either treatment arm, children will be provided with the medication, Albendazole will be given in syrup form, and Ivermectin tablet will be given in powdered form as Ivermectin suspension is not available in Bangladesh. Following all the aseptic procedure, the investigatorswill crush the commercially available 6 mg unscored Ivermectin tablets make a powder form with the tablet fragments, and preserve them in an airtight plastic container in a cool and dry place. According to the weight of the children, the investigators will provide the needed amount (weighted by microgram scale) of the drug mixed with 5 ml of water. Study fiield staffs will help the parents to give the medicine to the child by the direct observation therapy (DOT) method. The parents will be advised to bring the children on an empty stomach in the morning. Ivermectin will be given first, and a light snack will be provided 30 minutes after taking ivermectin. Then albendazole will be given to the children. Both drugs will be given using direct observation at the field clinic. Parents will be advised to report any adverse effects including vomiting, after taking medication. If vomiting occurs within one hour of medication, a redosing will be provided.

Blinding and procedures for unblinding This study will be an single blinded clinical trial. The investigators and study physicians will not be blinded. The investigators are not using any placebo arm for this trial, the approach to concealing the treatment arm by random selection of the study participants will avoid selection bias in the study. However, the primary objective of the study is a cure assessment of STH infection, which will be performed based on the egg reduction rate (ERR) with stool samples. To ensure the avoidance of any bias in the test, the laboratory personnel doing the procedures will be blinded.

Lab procedures:

Stool sample collection and microscopic examination: One fresh morning stool sample will be collected from each suspected STH-infected child at baseline and follow-up periods. The stool samples will be carried out to the field clinic within 30 minutes of collection, and slide preparation and other processing will be done in the next 30 minutes, and every sample should be assessed within one hour of the collection time. The expert field staffs and laboratory personnel will coordinate the entire process. Duplicate Kato-Katz thick smears will be prepared for each stool sample using 41.7 mg templates. All slides will be scrutinized within 60 minutes after preparation to prevent the over-clearing of hookworm eggs. To ensure the accuracy of microscopic diagnoses, 10% of the Kato-Katz thick smears will be randomly selected for a re-examination. In instances of conflicting results, slides will undergo a third reading, and the outcomes will be deliberated upon until a consensus is achieved; the agreement between the initial readings of the Kato-Katz thick smears and the quality control process should exceed 95%. In all the follow-up periods (five times) the same methods will be applied, so a total of six times stool samples will be collected from each child. At the field site, skilled and trained laboratory personnel will perform all laboratory investigations and examine thick smears for the presence of eggs from TT, hookworm, and AL during the enrolment and follow-up periods.

Blood: Only at baseline and 3 months follow-up, the investigatorswill also collect 2-4 ml of blood following all standard and aseptic techniques, using a butterfly needle for the child, which will puncture a vein in the elbow and blood will slowly suck into the syringe. After collecting blood, the needle will be pulled out gently and participants will be asked to continue to press the puncture site with alcohol cotton for a while until the bleeding stops, and then a band-aid will be applied to it. Then the collected blood will be assessed following all the standard procedures for slide preparation and cell counts for complete blood count (CBC) to evaluate anaemia and/or any other abnormalities.

Kato-Katz technique:

The cellophane faecal thick-smear examination (Kato-Katz technique) has proved to be an efficient means of diagnosis of soil-transmitted helminths. Cellophane thick-smear slides can be prepared in the field, stored in microscopic slide boxes, and shipped at great distances, for examination at a central laboratory if required. To ensure accurate and reliable results, quality control must be applied to laboratory procedures for diagnosing parasitic infections. Controls must apply to the collection of specimens, preparation of reagents, performance of the techniques, and examination of the final preparations.

The foundation of the Kato-Katz approach is a stool sample of variables (usually 41.7 mg) weighted using a sieved stool sample filled in a template hole. Therefore, it is necessary to apply a multiplication factor to convert the number of eggs observed by microscopy to EPG. The AM EPG of the two or four slides per participant will be calculated at baseline for each parasite species, study, and treatment group within the study if applicable.

Egg Reduction Rate (ERR) and Cure Rate (CR) Assessment Egg count assessments are usually longitudinal, which means that the same subjects are evaluated both before and after taking medication. In both medication trials and field settings, it is standard procedure to reject participants with zero pretreatment egg counts from additional testing to conserve resources.

Cure rate (CR) and egg reduction rate (ERR) are two typical ways to express drug efficacy. The WHO-recommended primary outcome measure for anthelmintic drug efficacy is the egg reduction rate (ERR). This quantitative measure expresses the percentage reduction in eggs per gram of stool (EPG) estimated before and after drug administration. The ERR is based on group arithmetic mean (AM) EPG, as recommended by WHO, rather than on individual EPG counts, however, the range of personal responses is broad.

The WHO-recommended reference efficacy standards are: "Anthelmintic drug efficacy is satisfactory if the ERR is superior or equal to the reference value; doubtful if the ERR is inferior to the reference value by less than 10 percentage points; reduced if the ERR is inferior to the reference value by at least 10 percentage points." The percentage of egg-positive people who turned egg-negative following treatment is known as the CR. Because CR requires no distributional assumptions and has a lower sensitivity to outliers than the ERR, it is frequently chosen for use in randomized clinical studies. However, in field settings, the ERR is preferable because it is more comparable across settings and is less impacted by pretreatment infection levels than the CR, which is lower at greater pretreatment egg counts.

ERR=[((meanEPG⁡count_(pre-treatment)-meanEPG⁡count_(post-treatment)))⁄(meanEPG⁡count_(pre-treatment) )]x100.

Individual ERR is calculated as the ratio of the difference between the pre-and post-treatment EPG to the pre-treatment EPG multiplied by one hundred. CRs and 95% binomial CIs were the percentage of stool-negative individuals at post-treatment follow-up. The distribution of individual responses in egg excretion was categorized as (i) negative (ERR = 100%, corresponding to the CR); (ii) reduction (ERR expressed as percentage reduction); (iii) no change or increase (ERR = 0), and further expressed in centiles.

Infection Intensity Classification:

The investigators will use the WHO-recommended cut-off values for analysing infection intensity at different follow-up periods based on faecal egg count found using the Kato-Katz technique.

Study Drug's labelling, and packaging Commercially available drugs will be used. Trial-specific labelling will be applied before use. icddr,b has a meticulous procurement policy and a strong procurement team. In case of unavailability of any drug, the investigators will procure the drug through the icddr,b logistics from any national and international pharmaceutical company. However, before purchasing the drug, the procurement team will assess the necessary documents, including the GMP certificate, certificate of analysis, and other regulatory documents from the respective companies. Only the drug satisfying the required standards will be obtained. All the drugs to be used in the study will be from a single source, and products from the same batch will be purchased to ensure the homogeneity of the drugs in terms of the quality and efficacy.

Accountability All study medications must be kept in a locked room that can be accessed only by the appropriate study personnel designated by the investigator. The study medications must not be used for other purposes other than this protocol. Under no circumstances may the investigator or site staff supply study medications to other investigators or sites or allow the medications to be used other than as directed by this protocol without prior authorization from the responsible party. Specific study forms for drug accountability will be designed to allow for adequate records on receipt, use, return, loss, or other medication disposition. The study pharmacist or designated personnel must maintain these accountability forms in a locked cabinet. Since the same drugs are used in routine practice, SOPs for labelling the boxes to be used in the trial will be developed, and the drugs used in the trial will be trial-specifically labelled and stored completely separated from the routine drugs. The compliance is assessed and reported in the CRF.

Storage Study drugs must be kept in a locked cabinet and/or in a room with restricted access, under the control of the experienced designated field staff. The temperature of the storage location will be monitored daily and recorded in a temperature log. In the event of temperature excursions below or above the allowable range, site staff must inform the study monitor. After testing the samples, the testing kits will be discarded using biohazard bags. The leftover samples will be stored in the icddr,b parasitology lab at -80* c temperature for 10 years. Samples will be discarded either after the storage period or if the parents don't allow the study team to store them for future use.

Concomitant treatments All medications required for concomitant conditions should be postponed until after the end of treatment for STH unless warranted by immediate medical need. Common conditions such as respiratory tract infections should be treated before starting treatment. There are no known interactions with other commonly used medications, though this cannot be excluded. All concomitant medications used during the study shall be recorded in the CRF. The investigators will also collect data if the children were given anti-helminthic drugs before or during the 6th, 9th, and 12th month follow-up by the guardians and physicians. In a randomized controlled trial, The investigators assume this can happen in both arms of the intervention, which will be analysed as mutually exclusive events in separate subgroups.

Safety & response to Treatment:

Safety: To ensure maximum patient safety, every patient will be physically examined (measuring height, weight, MUAC, general and systemic clinical examination etc.) before and during the follow-up period. The investigators will exclude patients with any abnormality, in addition to other conditions such as hypersensitivity to the study drugs, known chronic disease, or any other developmental abnormalities. All medications required for any other concurrent medical condition will be warranted for immediate treatment until STH infection treatment is completed. Treatment of common illnesses such as respiratory tract infections, will be ensured before STH medication is administered. The drug used in the study has no known interactions or risks with other commonly used drugs. The history of taking all other drugs used during the study will be recorded in the case report form. The investigators will monitor the children for any adverse events during treatment and follow-up, and guardians of the children will be advised to report any adverse events to the research team.

Response: Response to treatment will be assessed at the 3rd week, 3rd month, 6th month, 9th month, and 12th month since treatment. The cure will be assessed microscopically using the egg reduction rate measurement at the 3rd week, 3rd month, 6th month, 9th month, and 12th month since treatment compared to the baseline data. The cure rate (CR) of STH infection was defined as the percentage of the infected population negative for helminth eggs after anthelminthic treatment. The egg reduction rate (ERR) was defined as the percentage reduction in egg intensity as measured by eggs per gram of faeces after anthelminthic treatment.

In the 3rd week of follow-up, cure assessment, and egg reduction rate will be measured and if the results are not satisfactory for the proposed combination therapy, a standard regimen of treatment will be advised to the participants. The re-infection will be assessed at different time points (3rd,6th,9th,12th month). A 3rd month of infection will be considered as initial treatment with negative outcomes. Here, also the standard drug therapy will be advised for the research participants.

Adverse event follow-up All adverse events after baseline should be followed until those are resolved, the investigator assesses them as chronic or stable or the subject participation in the trial ends (i.e., until a final report is completed for that subject) . Guardian of the participant children will be advised to report any adverse event immediately after providing the medication to the child. The investigators will also collect data regarding any adverse event during each follow-up periods and document it in the case report form.

Quality Assurance:

According to the GCP, the investigators will implement and maintain quality assurance and quality control systems with written Standard Operating Procedures (SOPs). Quality control will be applied to each stage of data handling. The investigators will prepare and maintain adequate and accurate source documents to record all observations and other pertinent data for each patient who entered the study. During the study, the investigators will check that written informed consent has been obtained from all patients correctly and that data are recorded correctly and completely. Monitoring visits will be conducted according to the GCP guidelines and applicable local regulations. The PI/investigators will visit the site while participants are enrolled in the study at regular intervals according to the monitoring plan.

Sample size calculation:

N = 2× {z1-α +z1-β/(δ-δ0)}2 × s2 Here, N samples in each group Z1-α= 1.645 (when, α= 0.05) Z1-β= 0.845 (when, β= 0.80) δ (assumed difference in cure rate between two groups) = 20* δ0 (acceptable difference in cure rate between two groups) = 15 S (Standard deviation) = 10

*(Assumed cure rate of new treatment = 80%, Cure rate of the standard drug = 60%) Therefore, N clinical superiority= 2 x {(1.645+0.845)/ (20-15)}2 x 102 =49.6 =50 Considering an attrition rate of 10%, the calculated sample size is 50+5=55 per arm.

Given a 29.1% prevalence of TT and/or Hookworm infection among the target population, around 300 PSACs will be screened to get the desired sample size. The funding amount requested is sufficient to enroll and treat the number of subjects included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged within 2-5 years
* Height > 90 cm and Weight > 15 kg
* Both Stunted (The WHO-recommended height-for-age Z (HAZ) cut-off point is <-2 SD) and Healthy children (The WHO-recommended height-for-age Z (HAZ) cut-off point is >-1 SD)
* Confirmed case of STH having single/co-infection of TT/hookworm/AL
* Clinically healthy
* Not received any medications for STH within the last six months
* Guardians willing to let the children participate voluntarily through informed written consent

Exclusion Criteria:

* Non-compliance with any inclusion criteria
* Known severe allergies or adverse reactions to any of the study drugs
* Having any pre-existing chronic disease
* Recent participation in any clinical trials (within 1 year)
* Inability to comply with the study requirements, including follow-up visits and treatment adherence
* Guardians unwilling to let the children participate

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Through study completion, an average of 1 year
  The investigators will determine the safety of ivermectin and albendazole combination therapy for STH among preschool-age children (ages 2-5 years old) by assessing severe adverse events (SAEs) assessed by CTCAE v4.0. An adverse event will be defined as severe if it causes or contributes to the death or hospitalization for life-threatening conditions or results in persistent or significant disability or incapacity or a medically significant event. Any SAE occurrence for any child will be considered unsafe for that child.
Determine statistically significant effect of combination therapy | 3 weeks, 3 months, 6 months, 9 months, 12 months after baseline enrolment
  The investigators will determine whether the efficacy of ivermectin and albendazole combination therapy has a statistically significant effect (p < 0.05) on cure rates (CR) and egg reduction rates (ERR) compared to albendazole monotherapy.

SECONDARY OUTCOMES:
Determine statistically significant effect of combination therapy on patient's nutritional status based on z-scores | 3 months, 6 months, 9 months, 12 months after baseline enrolment
  The investigators will determine if Ivermectin and Albendazole combination therapy has a statistically significant effect (p < 0.05) on patients' nutritional status compared to Albendazole monotherapy. For that, the investigators will measure the height (in meters) and weight (in kilograms) of the children at baseline and in every follow-up period. Weight and height will be combined to report BMI in kg/m^2. The investigators will then calculate the z-scores for height and weight according to age of the children using WHO Anthro software, v3.2.2, Switzerland.
Correlate and compare changes in CR and ERR at different time points | 3 weeks, 3 months, 6 months, 9 months, 12 months after baseline enrolment
  The investigators will correlate and compare changes in CR and ERR at different time points and patient outcomes according to the types STH infection.
Determine statistically significant effect of combination therapy on patient's clinical condition (anaemia) based on haemoglobin count | At Baseline and 3 months after baseline enrolment
  The investigators will determine if Ivermectin and Albendazole combination therapy has a statistically significant effect (p < 0.05) on patients' clinical condition (anaemic status) compared to Albendazole monotherapy. For that, the investigators will conduct routine complete blood count (CBC) tests at baseline and 3-month follow-up periods and compare the mean of haemoglobin count and red cell indices (MCH, MCV, MCHC). Thus, evaluation of anemia will be used as an indicator of improvement of the clinical condition of the child.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Nazin Morshed, MBBS, Principal Investigator — International Centre for Diarrhoeal Diseases Research, Bangladesh (icddr,b)
Locations (1):
- International Centre for Diarrhoeal Diseases Research, Bangladesh (icddr,b), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pabalan N, Singian E, Tabangay L, Jarjanazi H, Boivin MJ, Ezeamama AE. Soil-transmitted helminth infection, loss of education and cognitive impairment in school-aged children: A systematic review and meta-analysis. PLoS Negl Trop Dis. 2018 Jan 12;12(1):e0005523. doi: 10.1371/journal.pntd.0005523. eCollection 2018 Jan. PMID 29329288
- [Background] Coulibaly YI, Dicko I, Keita M, Keita MM, Doumbia M, Daou A, Haidara FC, Sankare MH, Horton J, Whately-Smith C, Sow SO. A cluster randomized study of the safety of integrated treatment of trachoma and lymphatic filariasis in children and adults in Sikasso, Mali. PLoS Negl Trop Dis. 2013 May 9;7(5):e2221. doi: 10.1371/journal.pntd.0002221. Print 2013. PMID 23675549
- [Background] Davlin SL, Jones AH, Tahmina S, Kawsar AA, Joshi A, Zaman SI, Rahman MM, Morawski BM, Deming MS, Imtiaz R, Karim MJ. Soil-transmitted helminthiasis in four districts in Bangladesh: household cluster surveys of prevalence and intervention status. BMC Public Health. 2020 May 12;20(1):672. doi: 10.1186/s12889-020-08755-w. PMID 32397986
- [Background] Le B, Monteiro MAA, Amaral S, Wand H, Matthews A, Hii SF, Clarke NE, Arkell P, Yan J, Engelman D, Fancourt N, Fernandes JL, Steer A, Kaldor J, Traub R, Francis JR, Nery SV. The impact of ivermectin, diethylcarbamazine citrate, and albendazole mass drug administration on the prevalence of scabies and soil-transmitted helminths in school-aged children in three municipalities in Timor-Leste: a before-after assessment. Lancet Glob Health. 2023 Jun;11(6):e924-e932. doi: 10.1016/S2214-109X(23)00134-1. PMID 37202027
- [Background] Palmeirim MS, Hurlimann E, Knopp S, Speich B, Belizario V Jr, Joseph SA, Vaillant M, Olliaro P, Keiser J. Efficacy and safety of co-administered ivermectin plus albendazole for treating soil-transmitted helminths: A systematic review, meta-analysis and individual patient data analysis. PLoS Negl Trop Dis. 2018 Apr 27;12(4):e0006458. doi: 10.1371/journal.pntd.0006458. eCollection 2018 Apr. PMID 29702653
- [Background] Marti H, Haji HJ, Savioli L, Chwaya HM, Mgeni AF, Ameir JS, Hatz C. A comparative trial of a single-dose ivermectin versus three days of albendazole for treatment of Strongyloides stercoralis and other soil-transmitted helminth infections in children. Am J Trop Med Hyg. 1996 Nov;55(5):477-81. doi: 10.4269/ajtmh.1996.55.477. PMID 8940976
- [Background] Krotneva SP, Coffeng LE, Noma M, Zoure HG, Bakone L, Amazigo UV, de Vlas SJ, Stolk WA. African Program for Onchocerciasis Control 1995-2010: Impact of Annual Ivermectin Mass Treatment on Off-Target Infectious Diseases. PLoS Negl Trop Dis. 2015 Sep 24;9(9):e0004051. doi: 10.1371/journal.pntd.0004051. eCollection 2015. PMID 26401658
- [Background] Flohr C, Tuyen LN, Lewis S, Minh TT, Campbell J, Britton J, Williams H, Hien TT, Farrar J, Quinnell RJ. Low efficacy of mebendazole against hookworm in Vietnam: two randomized controlled trials. Am J Trop Med Hyg. 2007 Apr;76(4):732-6. PMID 17426180
- [Background] Lammie PJ, Fenwick A, Utzinger J. A blueprint for success: integration of neglected tropical disease control programmes. Trends Parasitol. 2006 Jul;22(7):313-21. doi: 10.1016/j.pt.2006.05.009. Epub 2006 May 19. PMID 16713738
- [Background] Awasthi S, Peto R, Pande VK, Fletcher RH, Read S, Bundy DA. Effects of deworming on malnourished preschool children in India: an open-labelled, cluster-randomized trial. PLoS Negl Trop Dis. 2008 Apr 16;2(4):e223. doi: 10.1371/journal.pntd.0000223. PMID 18414647
- [Background] Gerber DJF, Dhakal S, Islam MN, Al Kawsar A, Khair MA, Rahman MM, Karim MJ, Rahman MS, Aktaruzzaman MM, Tupps C, Stephens M, Emerson PM, Utzinger J, Vounatsou P. Distribution and treatment needs of soil-transmitted helminthiasis in Bangladesh: A Bayesian geostatistical analysis of 2017-2020 national survey data. PLoS Negl Trop Dis. 2023 Nov 6;17(11):e0011656. doi: 10.1371/journal.pntd.0011656. eCollection 2023 Nov. PMID 37930980
- [Background] Garg R, Lee LA, Beach MJ, Wamae CN, Ramakrishnan U, Deming MS. Evaluation of the Integrated Management of Childhood Illness guidelines for treatment of intestinal helminth infections among sick children aged 2-4 years in western Kenya. Trans R Soc Trop Med Hyg. 2002 Sep-Oct;96(5):543-8. doi: 10.1016/s0035-9203(02)90435-9. PMID 12474486
- [Background] Awasthi S, Verma T, Kotecha PV, Venkatesh V, Joshi V, Roy S. Prevalence and risk factors associated with worm infestation in pre-school children (6-23 months) in selected blocks of Uttar Pradesh and Jharkhand, India. Indian J Med Sci. 2008 Dec;62(12):484-91. PMID 19265242
- [Background] Brooker S, Kabatereine NB, Smith JL, Mupfasoni D, Mwanje MT, Ndayishimiye O, Lwambo NJ, Mbotha D, Karanja P, Mwandawiro C, Muchiri E, Clements AC, Bundy DA, Snow RW. An updated atlas of human helminth infections: the example of East Africa. Int J Health Geogr. 2009 Jul 9;8:42. doi: 10.1186/1476-072X-8-42. PMID 19589144
- [Background] Coffeng LE, Stolk WA, de Vlas SJ. Predicting the risk and speed of drug resistance emerging in soil-transmitted helminths during preventive chemotherapy. Nat Commun. 2024 Feb 6;15(1):1099. doi: 10.1038/s41467-024-45027-2. PMID 38321011
- [Background] Zeleke AJ, Bayih AG, Afework S, Gilleard JS. Treatment efficacy and re-infection rates of soil-transmitted helminths following mebendazole treatment in schoolchildren, Northwest Ethiopia. Trop Med Health. 2020 Nov 12;48(1):90. doi: 10.1186/s41182-020-00282-z. PMID 33292853
- [Background] Dunn JC, Bettis AA, Wyine NY, Lwin AMM, Tun A, Maung NS, Anderson RM. Soil-transmitted helminth reinfection four and six months after mass drug administration: results from the delta region of Myanmar. PLoS Negl Trop Dis. 2019 Feb 15;13(2):e0006591. doi: 10.1371/journal.pntd.0006591. eCollection 2019 Feb. PMID 30768602
- [Background] Prevalence of Soil Transmitted Helminths (STH) Infection among Children Aged 2-17 Years in Urban and Rural Areas of Dhaka District in Bangladesh
- [Background] Moser W, Schindler C, Keiser J. Efficacy of recommended drugs against soil transmitted helminths: systematic review and network meta-analysis. BMJ. 2017 Sep 25;358:j4307. doi: 10.1136/bmj.j4307. PMID 28947636
- [Background] WHO Expert Committee. Prevention and control of schistosomiasis and soil-transmitted helminthiasis. World Health Organ Tech Rep Ser. 2002;912:i-vi, 1-57, back cover. PMID 12592987
- [Background] Mekonnen Z, Hassen D, Debalke S, Tiruneh A, Asres Y, Chelkeba L, Zemene E, Belachew T. Soil-transmitted helminth infections and nutritional status of school children in government elementary schools in Jimma Town, Southwestern Ethiopia. SAGE Open Med. 2020 Sep 4;8:2050312120954696. doi: 10.1177/2050312120954696. eCollection 2020. PMID 32953118
- [Background] Dhakal S, Karim MJ, Al Kawsar A, Irish J, Rahman M, Tupps C, Kabir A, Imtiaz R. Post-intervention epidemiology of STH in Bangladesh: Data to sustain the gains. PLoS Negl Trop Dis. 2020 Dec 7;14(12):e0008597. doi: 10.1371/journal.pntd.0008597. eCollection 2020 Dec. PMID 33284834
- [Background] Neglected Tropical Diseases in Bangladesh: Situation Analysis and Gap Analysis. Dhaka; 2011.
- [Background] Edoa JR, Adegbite BR, Honkpehedji YJ, Zinsou JF, Boussougou-Sambe ST, Woldearegai TG, Mordmuller B, Adegnika AA, Dejon-Agobe JC. Epidemiology of soil-transmitted helminth infections and the differential effect of treatment on the distribution of helminth species in rural areas of Gabon. Trop Med Health. 2024 Jan 2;52(1):3. doi: 10.1186/s41182-023-00567-z. PMID 38163912
- See also: World Health Organization (WHO). Neglected tropical diseases — https://www.who.int/news-room/questions-and-answers/item/neglected-tropical-diseases
- See also: Children Without Worms (CWW) — https://childrenwithoutworms.org/about-sth/%0A
- See also: Organization WH. Soil-transmitted helminthiases: eliminating as public health problem soil-transmitted helminthiases in children: progress report 2001-2010 and strategic plan 2011-2020 — https://iris.who.int/handle/10665/44804
- See also: Organization WH. 2030 targets soil-transmitted helminthiases control programs — https://iris.who.int/handle/10665/330611